CLINICAL TRIAL: NCT03409289
Title: (RHAPSody) Diagnostic Utility of the Rapid Ultrasound for Shock and Hypotension (RUSH) Exam Following Return of Spontaneous Circulation (ROSC) in Cardiac Arrest
Brief Title: RHAPSody: Diagnostic Utility of RUSH Following ROSC
Status: Terminated | Type: Observational
Why Stopped: Expired IRB
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201702314; OCR18537 (Other: University of Florida)
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Cardiac Arrest
Keywords: Spontaneous Circulation (ROSC); Shock and Hypotension (RUSH) exam
MeSH Terms: conditions — Heart Arrest; Shock; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- ROSC RUSH Exam: The study population will include out of hospital cardiac arrest (both traumatic and non-traumatic causes) with return of spontaneous circulation after the cardiac arrest while in the emergency department .
  Interventions: Device: RUSH Exam

INTERVENTIONS:
Device: RUSH Exam — Within two hours of return of spontaneous circulation, the following elements of the RUSH exam will be performed: focused evaluation of the heart, inferior vena cava, abdomen and aorta with the addition of evaluation for DVT and ocular ultrasound.

SUMMARY:
This will be a prospective observational study of adult primary cardiac arrest patients presenting to Shands Emergency Department following ROSC or actively in cardiac arrest with subsequent ROSC after treatment in the emergency department.

DETAILED DESCRIPTION:
This will be a prospective observational study of adult primary cardiac arrest patients presenting to Shands Emergency Department following ROSC or actively in cardiac arrest with subsequent ROSC after treatment in the emergency department. The study will be a single center pilot study to evaluate the role of the extended RUSH exam in patients following cardiac arrest in order to potentially diagnose the cause of their arrest. No control group will be included in this study due to ethical concerns of withholding a potentially life-saving diagnostic test. Patients will be treated with ACLS per standard of care and resuscitation measures given. Within two hours of return of spontaneous circulation, the RUSH exam will be performed by ultrasound-trained emergency department physicians with images saved into the Qpath system, our already existing database where all emergency ultrasound exams - education and diagnostic - are stored currently. The physician who performed the exam will fill out a checklist with their interpretation and findings based on the elements included in the exam. The data collected will be stored in a RedCap database. Identifying data will be removed from the images and reviewed by two experienced ultrasonographers who will give separate interpretations, and inter-observer reliability will be examined. We will then correlate the interpretation with that of the physicians performing the exam. The elements of the RUSH exam that will be performed include focused evaluation of the heart, inferior vena cava, abdomen and aorta with the addition of evaluation for DVT and ocular ultrasound. The evaluation for DVT will be an abbreviated exam with one view of each of the bilateral femoral veins and popliteal veins. Techniques for performing the exam are based on the 2012 RUSH guidelines [2]. The data will undergo statistical analysis to determine if the data supported the initial hypotheses. Subjects will be contacted 30 days following the initial study for telephone follow-up and a CPC assessment for neurologic recovery will also be performed at that time.

ELIGIBILITY:
Inclusion Criteria:

* Incoming ER patients with return of spontaneous circulation after cardiac arrest

Exclusion Criteria:

* Patients who do not achieve return of spontaneous circulation long enough for the exam to be performed
* Patients who have initial cardiac arrest while on an inpatient unit of the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute care adult patients with cardiac arrest, including both traumatic and non-traumatic causes.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Cause of cardiac arrest. | length of hospital stay (7 days)
  Assessment of a contributing diagnosis or cause of cardiac arrest following performance of the extended RUSH exam. We will examine if a diagnosis is provided or supported by the RUSH exam and if this leads to intervention.

SECONDARY OUTCOMES:
Intervention or treatment initiated based on the results of the exam | length of hospital stay (7 days)
  Shorten time to critical interventions and/or treatment
Time to ultimate diagnosis (if found) | length of hospital stay(7 days)
  Shorten length of time from presentation at ER to ultimate diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie C. Nickels, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health (UFHealth), Gainesville, Florida, United States